CLINICAL TRIAL: NCT00221299
Title: Can Risedronate and Parathyroid Hormone Reverse Glucocorticoid Induced Osteoporosis?
Brief Title: Risedronate and Parathyroid Hormone to Reverse Osteoporosis Caused by Chronic Steroid Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Nancy E. Lane, MD, Principal Investigator, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200513216
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Steroids; Prednisone
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid; Parathyroid Hormone; Teriparatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group1a-rhPTH&RIS-Placebo(Y1)&RIS(Y2) (Active Comparator): First phase (year 1) - parathyroid hormone (rhPTH 1-34), 20 ug SC injections daily and risedronate placebo tablets for one year Second phase (year 2) - re-randomized to risedronate (35mg/wk) tablets for second year.
  Interventions: Drug: Risedronate; Drug: Parathyroid Hormone
- Group1b-rhPTH&RisendronatePlacebo (Active Comparator): First phase (year 1) - parathyroid hormone (rhPTH 1-34), 20 ug SC injections daily and risedronate placebo tablets for one year Second phase (year 2) - continue on risedronate placebo tablets for second year.
  Interventions: Drug: Parathyroid Hormone
- Group2-rhPTH&Risedronate (Active Comparator): First phase (year 1) - parathyroid hormone (rhPTH 1-34), 20 ug SC injections daily and risedronate tablets (35mg/wk) tablets for one year Second phase (year 2) - continue on risedronate tablets (35mg/wk) for second year.
  Interventions: Drug: Risedronate; Drug: Parathyroid Hormone
- Group3-rhPTH-Placebo&Risedronate (Active Comparator): First phase (year 1) - parathyroid hormone (rhPTH 1-34), placebo SC injections of normal saline daily and risedronate tablets (35mg/wk) tablets for one year Second phase (year 2) - continue on risedronate tablets (35mg/wk) for second year.
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate — One 35mg tab of risedronate/placebo taken once a week for one year.
  Other Names: Actonel, NDC# 0149-0472-04
  Arms: Group1a-rhPTH&RIS-Placebo(Y1)&RIS(Y2); Group2-rhPTH&Risedronate; Group3-rhPTH-Placebo&Risedronate
Drug: Parathyroid Hormone — This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
  Other Names: Forteo; PTH; rhPTH 1-34; NDC# 0002-8971-01
  Arms: Group1a-rhPTH&RIS-Placebo(Y1)&RIS(Y2); Group1b-rhPTH&RisendronatePlacebo; Group2-rhPTH&Risedronate

SUMMARY:
The purpose of the study is to learn if one year of treatment with parathyroid hormone (PTH), either alone or with risedronate, will increase the thickness of the bones in the hip and spine in subjects with osteoporosis from chronic low dose steroid use. During the second year, the study will also look at whether taking risedronate will preserve the bone thickness created by one year of rhPTH 1-34 treatment.

DETAILED DESCRIPTION:
Dr. Nancy Lane and colleagues at the University of California, Davis and University of California, San Francisco will be conducting this 2-year study of human parathyroid hormone (rhPTH 1-34) alone, and rhPTH (1-34) with risedronate compared to risedronate alone in men and women with osteopenia on chronic low dose glucocorticoids (GC). This is an investigator-initiated study funded by Aventis Pharmaceuticals.

The study will be divided into 2 phases. All study subjects will receive supplemental calcium citrate and Vitamin D during the 2-year study. In year one subjects will be randomly assigned to receive PTH (subcutaneously daily) or placebo and risedronate tablets or placebo. In year two, PTH will be stopped and subjects in group 1 will be re-randomized to receive risedronate tablets or placebo. Subjects in group 2 and 3 will continue on risedronate tablets.

In year one of the study, subjects were randomly assigned to one of the following treatment groups.

1. Group 1: rhPTH (1-34) (20ug subcutaneously daily) + riesdronate placebo tablets
2. Group 2: rhPTh (1-34) (20ug subcutaneously daily) + risedronate tablets (35mg/wk)
3. Group 3: rhPTh placebo (subcutaneous injections of normal saline) + risedronate tablets (35mg/wk)

In year two of the study, beginning at the 12 month timepoint

1. Group 1 subjects were re-randomized to either:

   Group 1a: risedronate (35mg/wk) or Group 1b: risedronate placebo
2. Group 2 subjects continued risedronate (35mg/wk)
3. Group 3 subjects continued risedronate (35mg/wk)

Potential study subjects will have dual x-ray absorptiometry measurements (DEXA) of the spine and hip at the screening visit. Those study subjects who meet the inclusion criteria will be invited back for a baseline visit.

DEXA scans of the spine, hip, and forearm will be done at Baseline visit, 6-month, 12-month, 18-month, and 24-month follow-up visits. DEXA scan of the spine, hip, and forearm takes approximately 20 minutes to complete. To assess incident vertebral and non-vertebral fractures, lateral thoracic and lumbar spine evaluation using Instant Vertebral Assessment [IVA] will be done at Baseline, 12-month, and 24-month follow-up visits.

The specific aims of the study are as follows:

1. To determine if changes in bone mineral density in the spine and hip caused by 1 year of treatment with rhPTH (1-34) alone then followed by risedronate or rhPTH (1-34) with risedronate are greater than PTH placebo and risedronate in patients with GIO who are taking calcium, MVIs and chronic low doses of glucocorticoids.
2. To determine if risedronate will preserve the high bone mass state created by 1 year of rhPTH (1-34) treatment.
3. To determine the association of biochemical markers of bone turnover with rhPTH (1-34) and risedronate both during and after treatment.
4. To compare, as possible, the fracture incidence between the rhPTH (1-34) alone followed by risedronate, and rhPTH (1-34) with risedronate compared to risedronate + placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, greater than 18 years of age with a history of glucocorticoid therapy with prednisone ≥ 7.5mg/d for 6 months, and currently on prednisone ≥ 5mg /day.
* DXA of the lumbar spine (L1-L4) or total hip or femoral neck T score ≤ -1.5 with or without a prevalent vertebral fracture. (The T score is the number of standard deviations above or below the population mean for young, normal pre-menopausal females age 30).
* Investigators are satisfied that that there is no physical condition that would prevent a patient from receiving the proposed treatment regimens.
* Patient is ambulatory and able to return to the site of the investigation at specified time during the study.
* The patient is willing to participate in the proposed study as evidenced by signing an informed consent.
* Women of childbearing age are willing to use 2 forms of contraception during the entire study period.
* Have at least one analyzable BMD site: lumbar spine and/or proximal femur

Exclusion Criteria:

* Generalized disease of bone other than related to a rheumatic disease and glucocorticoid-induced osteoporosis including: hyperparathyroidism, hypoparathyroidism, Paget's disease of bone
* Diseases that may affect bone metabolism including: alcoholism, hyperthyroidism, renal impairment (creatinine > 2.5mg/dl) or hepatic impairment (SGOT levels > 2x upper limit of normal
* Urinary excretion of calcium > 400mg/day
* History of drug abuse
* Previous use of alendronate within 6 months prior to the study
* Previous use of risedronate, hormone replacement therapy or calcitonin within 2 months prior to the study
* History of unstable cardiovascular disease or uncontrolled hypertension
* Severe scoliosis, greater than 2 lumbar fractures, or spinal surgery such that a precise bone mass measurement could be affected
* History of gastrointestinal intolerance to bisphosphonates
* History of cancer within 5 years of the study
* Patients on glucocorticoids for organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Lane, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis General Medicine Research Clinic, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group1a-rhPTH&RIS-Placebo(Y1)&RIS(Y2): First phase (year 1) - parathyroid hormone (rhPTH 1-34), 20 ug SC injections daily and risedronate placebo tablets for one year Second phase (year 2) - re-randomized to risedronate (35mg/wk) tablets for second year.
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for year 1. One 35mg tab of risedronate taken once a week for year 2.
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Group1b-rhPTH&RisendronatePlacebo: First phase (year 1) - parathyroid hormone (rhPTH 1-34), 20 ug SC injections daily and risedronate placebo tablets for one year Second phase (year 2) - continue on risedronate placebo tablets for second year.
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for two years.
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Group2-rhPTH&Risedronate: First phase (year 1) - parathyroid hormone (rhPTH 1-34), 20 ug SC injections daily and risedronate tablets (35mg/wk) tablets for one year Second phase (year 2) - continue on risedronate tablets (35mg/wk) for second year.
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for two years.
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Group3-rhPTH-Placebo&Risedronate: First phase (year 1) - parathyroid hormone (rhPTH 1-34), placebo SC injections of normal saline daily and risedronate tablets (35mg/wk) tablets for one year Second phase (year 2) - continue on risedronate tablets (35mg/wk) for second year.
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for two years.
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
Period: Overall Study
Arm/Group | Group1a-rhPTH&RIS-Placebo(Y1)&RIS(Y2) | Group1b-rhPTH&RisendronatePlacebo | Group2-rhPTH&Risedronate | Group3-rhPTH-Placebo&Risedronate
Started | 11 | 13 | 14 | 11
Completed | 10 | 11 | 14 | 10
Not Completed | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study subjects were men and women, greater than 18 years of age with a history of glucocorticoid therapy with prednisone >= 7.5gm a day for 6 months and currently on prednisone or equivalent >= 5mg/day.
Groups:
- Parathyroid Hormone Injections and Risedronate Placebo Tablets: parathyroid hormone (rhPTH 1-34) injections and risedronate placebo tablets for one year
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Parathyroid Hormone Injections and Risedronate Tablets: Parathyroid hormone (rhPTH 1-34) injections and risedronate tablets for one year
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for one year.
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Parathyroid Hormone Placebo Injections and Risedronate Tables: parathyroid hormone (rhPTH 1-34) placebo injections and risedronate tablets for one year
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for one year.
- Total: Total of all reporting groups
Arm/Group | Parathyroid Hormone Injections and Risedronate Placebo Tablets | Parathyroid Hormone Injections and Risedronate Tablets | Parathyroid Hormone Placebo Injections and Risedronate Tables | Total
Number analyzed (Participants) | 24 | 14 | 11 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (14) | 48.3 (14.9) | 53 (18.8) | 50.6 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 14 | 11 | 49
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 14 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD): Examine the Pattern and Effect of BMD Changes at Hip and Spine Measured by DXA Every 6 Months.
Description: In this randomized clinical trial to determine if treatment with rhPTH (1-34) with and without risedronate will increase bone mass of the lumbar spine more than risedronate alone. This was a small pilot study and study subjects were recruited from two study sites. Our primary endpoint was change in lumbar spine BMD.
Time Frame: BMD changes from year 1 to year 2
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Parathyroid Hormone&Risedronate Placebo: parathyroid hormone (rhPTH 1-34) injections and risedronate placebo tablets for one year
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Parathyroid Hormone&Risedronate: Parathyroid hormone (rhPTH 1-34) injections and risedronate tablets for one year
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for one year.
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Parathyroid Hormone Placebo&Risedronate: parathyroid hormone (rhPTH 1-34) placebo injections and risedronate tablets for one year
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for one year.
Arm/Group | Parathyroid Hormone&Risedronate Placebo | Parathyroid Hormone&Risedronate | Parathyroid Hormone Placebo&Risedronate
Number analyzed (Participants) | 21 | 14 | 10
percent change | 0.85 (0.10) | 0.84 (0.12) | 0.91 (0.11)

ADVERSE EVENTS:
Description: Serious and/or other (non-serious) adverse events were collected/assessed, but none observed.
Groups:
- Parthyroid Hormone Injections and Risedronte Tablets: Parathyroid hormone (rhPTH 1-34) injections and risedronate tablets for one year
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for one year.
  Parathyroid Hormone: This medication comes in a pre packaged 28 day supply pen. Medication is administered once a day by a subcutaneous injection (under the skin) into the thigh or abdomen. For this study, this medication will be taken for one year.
- Parathyroid Hormone Placebo Injections and Risedronate Tablets: parathyroid hormone (rhPTH 1-34) placebo injections and risedronate tablets for one year
  Risedronate: One 35mg tab of risedronate/placebo taken once a week for one year.
Arm/Group | Parathyroid Hormone Injections and Risedronate Placebo Tablets | Parthyroid Hormone Injections and Risedronte Tablets | Parathyroid Hormone Placebo Injections and Risedronate Tablets
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/24 | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No